CLINICAL TRIAL: NCT05010538
Title: A Single Center, Phase 4, Open-label Prospective Case Series Study of the Safety and Efficacy of Sarecycline for 12 Weeks in Subjects Ages 9 and Over With Truncal Acne
Brief Title: Sarecycline Truncal Acne Safety and Efficacy Response
Acronym: TASER
Status: Completed | Type: Observational
Sponsor: Angela Moore (Other)
Collaborators: Almirall, SAS (Industry)
Responsible Party: Sponsor-Investigator, Angela Moore, Principal Investigator, Arlington Research Center
Organization: Arlington Research Center (Other)
Other Study IDs: Sarecycline TASER1
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Sarecycline; Tetracycline; Truncal Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — sarecycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sarecycline: Eligible patients will be prescribed with commercially available sarecycline at a dosage of 1.5 mg/kg/day and followed for 12 weeks post initiation of treatment.
  Interventions: Drug: Sarecycline

INTERVENTIONS:
Drug: Sarecycline — 60 mg sarecycline tablets will be given for subjects with a body weight of 33 to 54 kg, 100 mg sarecycline tablets will be given for subjects with a body weight of 55 to 84 kg, and 150 mg tablets will be given for subjects with a body weight between 85 and 136 kg.
  Other Names: Seysara®

SUMMARY:
The purpose of this study is to determine the efficacy and safety of oral sarecycline 1.5 mg/kg/day in truncal acne. Patients with moderate to severe acne vulgaris will be observed over a period of 12 weeks. Lesion counts, investigator's global assessments, photography, and safety measures will be assessed for the trunk and face.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 9 or above.
* Clinical diagnosis of moderate to severe truncal acne based on IGA

Exclusion Criteria:

* Known or suspected allergies or sensitivities to any components of the study drug.
* Any disorders that would preclude the use of tetracycline-class antibiotics or sarecycline.
* Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with the interpretation of the trial results and/or put the subject at significant risk (according to the Investigator's judgment) if the subject takes part in the trial.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 9 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with moderate to severe truncal acne at a single center in Texas, USA.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Acne Severity Based on Investigator's Global Assessment Success | Baseline, Week 12
  Investigator's Global Assessment (IGA) success for truncal acne vulgaris at week 12
Change from Baseline in Absolute Lesion Count | Baseline, Week 12
  Absolute change from baseline lesion counts for inflammatory acne for truncal acne vulgaris at week 12

SECONDARY OUTCOMES:
Adverse Events and Adverse Events of Special Interest | Baseline, Week 12
  Safety based on adverse events (AEs), adverse events of special interest (AESI), vital signs, and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Angela Moore, MD, Principal Investigator — Arlington Research Center
Locations (1):
- Arlington Research Center, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No